CLINICAL TRIAL: NCT01853293
Title: Use of Kudzu Extract in the Study of Its Ability to Reduce Alcohol Drinking in Treatment Seeking Alcohol Dependent Persons
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Grant was not funded
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, David M. Penetar, Psychologist, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-000727
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Alcohol Abuse; Alcohol Dependence; Heavy Drinking Days
Keywords: Alcohol Abuse; Alcohol Dependence; Heavy drinking days; Kudzu
MeSH Terms: conditions — Alcoholism | interventions — Practice Management, Medical

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kudzu extract (Active Comparator): Participants will take two 500-mg capsules of Kudzu extract, t.i.d. (morning, 6:00 to 8:30 a.m.; afternoon, 2:00 to 4:30 p.m.; evening, 9:00 to 11:30 p.m.).
  Interventions: Drug: Kudzu extract; Behavioral: Medical Management
- Placebo (Placebo Comparator): Placebo capsule contains sugar beet filler. Participants will take two 500-mg capsules, t.i.d. (morning, 6:00 to 8:30 a.m.; afternoon, 2:00 to 4:30 p.m.; evening, 9:00 to 11:30 p.m.).
  Interventions: Drug: Placebo; Behavioral: Medical Management

INTERVENTIONS:
Drug: Kudzu extract
  Arms: Kudzu extract
Drug: Placebo
  Arms: Placebo
Behavioral: Medical Management — Medical Management is a manualized treatment deriving from a number of empirically tested manualized therapies designed to approximate a primary care approach to alcohol dependence. The treatment, delivered by a medical professional (i.e., nurse or physician), monitors medication side effects, provides strategies to increase medication adherence and supports abstinence through psychoeducation and referral to groups such as Alcoholics Anonymous. The visits allow for assessments of drinking, overall functioning, medication adherence, and side effects. Also at one of these weekly visits, a blood sample will be taken for liver function tests (GGT, ALT, AST). Samples will be further analyzed for two measures of heavy drinking: carbohydrate deficient transferrin (CDT) and phosphatidylethanol (PEth).

SUMMARY:
This research is designed to assess if problem drinking by treatment seeking individuals can be treated (reduced) by kudzu extract pharmacotherapy plus medical management therapy.

DETAILED DESCRIPTION:
Men and women participants, ages 21-60 yrs old and seeking treatment for their drinking, but otherwise physically and mentally healthy, will be recruited. Participants must meet criteria for heavy drinking* and either Alcohol Abuse or Alcohol Dependence according to DSM-IV criteria. Following a baseline period, participants will be randomized to take either kudzu extract or placebo for 10 weeks, and record and report their alcohol consumption. All participants will receive weekly medical management sessions with the study physician.

*Heavy Drinking according to the National Institute on Alcohol Abuse and Alcoholism (2007) is more than 4 drinks per day and more than 14 drinks per week for men; and for women, more than 3 drinks per day and more than 7 drinks per week.

ELIGIBILITY:
Inclusion Criteria:

* Treatment seeking for alcohol abuse or dependence.
* Non cigarette smokers are preferred, but will accept those who smoke less than 10 cigarettes per day.
* Marijuana use of less than once per week. Other drug use less than 20 lifetime uses.
* Absence of current Axis I disorders except alcohol abuse or dependence. Past diagnosis (greater than 1 year) is acceptable.
* BMI within 18-30.
* Physically healthy (normal physical exam, ECG, blood and urine chemistries).
* Female participants must use medically approved method of contraception. If barrier method is used, must agree to using two methods simultaneously (e.g., diaphragm and condom).

Exclusion Criteria:

* Taking any prescription medication (except oral contraceptives, certain short term anti -fungal agents and some topical creams for dermal conditions).
* On psychotropic medications.
* Drug use (other than nicotine, alcohol or marijuana) greater than 20 lifetime uses.
* Meets criteria for current drug abuse or dependence (other than alcohol and nicotine). Past abuse/dependence (greater than 3 years) is acceptable.
* History of major head trauma.
* History of cardiac problems.
* Pregnancy, lactating, or planning to become pregnant during the study period.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Percentage of heavy drinking days | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David M. Penetar, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Behavioral Psychopharmacology Research Laboratory, Belmont, Massachusetts, United States